CLINICAL TRIAL: NCT03353155
Title: Can Refinements to Effective Transitional Care Services Improve Outcomes? Results From a Pragmatic, Randomized Controlled Trial.
Brief Title: Effectiveness of Transitional Care Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National University Health System, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NUHSCareHub
Record Dates: First submitted 2017-11-12; First posted 2017-11-27 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Post-cardiac Surgery

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned to one of two groups. Group 1 is usual care, in which patients are followed up after surgery by the ambulatory clinic assigned to their case. Patients in usual care have access to occupational and physical therapy, and medical social work, if they choose to use them. Group 2 is CareHub, in which patients are followed up by a dedicated care coordinator who proactively calls patients at home and schedules their clinic appointments, and consults with therapists and medical social workers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Telephone and/or home visits at 1 week, and thereafter, monthly for 6 months, to check on medication compliance and/or medical social problems and/or physical therapy needs and/or health-related financial challenges by the relevant service departments as recommended by the discharging physician.
  Interventions: Behavioral: Usual Care
- CareHub (Active Comparator): Telephone follow-up by a nurse care coordinator acting as single point of contact for medication compliance and/or medical social problems and/or physical therapy needs and/or health-related financial challenges based on automatic enrollment using ACE score cut-off at admission.
  Interventions: Behavioral: CareHub

INTERVENTIONS:
Behavioral: Usual Care
  Arms: Usual Care
Behavioral: CareHub
  Arms: CareHub

SUMMARY:
The National University Hospital System has designed and is piloting an improved post-discharge care programme called CareHub for patients undergoing cardiac surgery. CareHub is a post-discharge care programme that is designed to streamline and better coordinate current programmes for patients at high risk of readmission.

To assess the clinical and cost-effectiveness of CareHub, our team will randomly assign patients to a usual care setting or CareHub setting, and measure clinical outcomes, patient satisfaction, readmissions, and length of stay through 6 months post-discharge in both groups.Patients enrolled in both groups will receive post-discharge care for six months after discharge. CareHub patients will receive a single point of contact for access to usual care services. Recruitment for this pilot will be from 20 April 2016 - approximately late October 2016, and the CareHub team will provide 6 months of post-discharge support. The entire pilot will thus run from 20 April 2016 - April / May 2017, with data collection extending 6 months after the last patient is enrolled.

DETAILED DESCRIPTION:
Today, the National University Hospital System has a variety of transitional / post-discharge care programmes, and patients may be enrolled in more than one. Each of these programmes is run by a different hospital team, so a patient may have to liaise with many parties for their post-discharge care.

The National University Hospital System has designed and is piloting an improved post-discharge care programme called CareHub for patients undergoing cardiac surgery. Recruitment for this pilot will be from 20 April 2016 - approximately late October 2016, and the CareHub team will provide 6 months of post-discharge support. The entire pilot will thus run from 20 April 2016 - April / May 2017.

CareHub is a post-discharge care programme that is designed to streamline and better coordinate current programmes for patients at high risk of readmission. Patients enrolled in CareHub and usual care will receive post-discharge care for six months after discharge. However, patients in CareHub will experience:

(i) Provision of a single point of contact for all the patient's needs, to help patients and their families navigate the healthcare system as well as various programmes available in the hospital and community. Care Coordinator identifies patients and starts working with care team during the inpatient phase, and follows patient through to the post-discharge phase.

(ii) More structured and regular telephone support and checks, to help ease the hospital-to-home transition, as well as to provide more opportunity to verify that patients are adhering to their recommended treatment (which may include e.g. checking that patients have made use of the daycare services CareHub recommended).

(iii) A call center which will operate during office hours, where tele-consult will be available from and nurses/care coordinators.

(iv) A consolidated multi-disciplinary discharge plan, based on the input of all healthcare workers caring for the patient. These include the CareHub coordinator, ward doctor and nurse, heart failure care manager, and allied health professionals, as required.

(v) Early identification and preparation for post-discharge care. Healthcare workers listed in (iv) will participate in a daily in-patient multi-disciplinary ward huddle, to discuss the patient's condition and start early preparation for post-discharge care.

To assess the clinical and cost-effectiveness of CareHub, our team will randomly assign patients to a usual care setting or CareHub setting, and measure clinical outcomes, patient satisfaction, readmissions, and length of stay through 6 months post-discharge in both groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the cardiac inpatient service post-cardiac surgery

Exclusion Criteria:

* Patients that do not consent or are unable to consent to be included into CareHub

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Post-discharge length of stay | 6 months
  Patient's length of stay for any readmissions following index admission
Unplanned readmissions | 6 months
  Whether patients were admitted for a cardiac complaint after index admission
Cardiac-related specialist outpatient clinic visits | 6 months
  The number of post-index admission visits to an outpatient clinic for cardiac consults
Emergency department visits | 6 months
  The number of emergency department visits post-index admission

SECONDARY OUTCOMES:
Net cost of service utilization | 6 months
  CareHub cost/patient minus Usual Care cost/patient

CONTACTS AND LOCATIONS:
Overall Officials: John Wong, MD, PhD, Principal Investigator — National University Hospital System; Phillip Phan, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participate data has been de-identified. There are currently no plans to share the data.

REFERENCES:
- [Background] Jencks SF, Williams MV, Coleman EA. Rehospitalizations among patients in the Medicare fee-for-service program. N Engl J Med. 2009 Apr 2;360(14):1418-28. doi: 10.1056/NEJMsa0803563. PMID 19339721
- [Background] Coleman EA. Falling through the cracks: challenges and opportunities for improving transitional care for persons with continuous complex care needs. J Am Geriatr Soc. 2003 Apr;51(4):549-55. doi: 10.1046/j.1532-5415.2003.51185.x. PMID 12657078
- [Background] Greysen SR, Harrison JD, Kripalani S, Vasilevskis E, Robinson E, Metlay J, Schnipper JL, Meltzer D, Sehgal N, Ruhnke GW, Williams MV, Auerbach AD. Understanding patient-centred readmission factors: a multi-site, mixed-methods study. BMJ Qual Saf. 2017 Jan;26(1):33-41. doi: 10.1136/bmjqs-2015-004570. Epub 2016 Jan 14. PMID 26769841
- [Background] Wee SL, Loke CK, Liang C, Ganesan G, Wong LM, Cheah J. Effectiveness of a national transitional care program in reducing acute care use. J Am Geriatr Soc. 2014 Apr;62(4):747-53. doi: 10.1111/jgs.12750. Epub 2014 Mar 17. PMID 24635373
- [Background] Coleman EA, Smith JD, Frank JC, Min SJ, Parry C, Kramer AM. Preparing patients and caregivers to participate in care delivered across settings: the Care Transitions Intervention. J Am Geriatr Soc. 2004 Nov;52(11):1817-25. doi: 10.1111/j.1532-5415.2004.52504.x. PMID 15507057
- [Background] Naylor M, Brooten D, Jones R, Lavizzo-Mourey R, Mezey M, Pauly M. Comprehensive discharge planning for the hospitalized elderly. A randomized clinical trial. Ann Intern Med. 1994 Jun 15;120(12):999-1006. doi: 10.7326/0003-4819-120-12-199406150-00005. PMID 8185149
- [Background] Allen J, Hutchinson AM, Brown R, Livingston PM. Quality care outcomes following transitional care interventions for older people from hospital to home: a systematic review. BMC Health Serv Res. 2014 Aug 15;14:346. doi: 10.1186/1472-6963-14-346. PMID 25128468

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT03353155/Prot_SAP_001.pdf